CLINICAL TRIAL: NCT01294501
Title: Decreasing Medication Errors by Caregivers Using a Health Literacy Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAI0786
Record Dates: First submitted 2011-02-04; First posted 2011-02-11 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Medication Administration; Medication Errors
Keywords: Medication administration; Medication errors; Health Literacy; Pediatric Emergency Department; Web-based education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fever assessment and management (Experimental): Medication administration educational module for low literacy subjects on how to administer common medications appropriately and safely.
  Interventions: Other: Medication administration educational module

INTERVENTIONS:
Other: Medication administration educational module — The Research Assistant (RA) will enter the subject's language (English or Spanish), the type of medicine (tablet/capsule, liquid, or ointment) from the antibiotic prescription, and the frequency (once a day, twice a day, three times a day, four times a day) from the antibiotic prescription into the web-based educational module on medication administration so that a tailored module will be setup for the subject. The subject will then view the educational interactive module. After the subject is done with the module, the RA will administer a verbal post-test. The post-test will include questions on medication administration as well as questions on fever assessment and management.
  Other Names: Health Literacy Intervention

SUMMARY:
Giving medications to children can be confusing; studies have shown that caregivers make dosing administration errors up to 50% of the time. There are many reasons that there are so many errors, including the fact that dosing for children is based on their weight, liquid medications come in many different forms, and caregivers often give medicines using kitchen teaspoons and tablespoons. Caregivers who have difficulty reading have even more difficulty understanding medication instructions. We are developing and testing a web-based educational module to teach caregivers how to give medications. We are focusing on the pediatric emergency department because we know that this population has low literacy levels, and that many antibiotics are prescribed in this setting. We anticipate that those caregivers that view the interactive module will have increased knowledge on how to give medications once they get home.

DETAILED DESCRIPTION:
Dosing error rates of home administration of medications to children have been reported to be as high as 50%. Contributing to this error rate are the complexity of pediatric weight-based dosing, confusing formulations of liquid medications, and a reliance on non-standardized dosing tools such as kitchen teaspoons and tablespoons to administer medications. Families with low health literacy are at particular risk for medication administration errors. Health literacy promoting interventions to improve medication administration such as dissemination of a pictogram-based medication list have been shown to work for common over-the-counter medications such as acetaminophen, but their effect on administration practices for common medications prescribed in the pediatric emergency department (PED) has not been evaluated. Of the 50,000 patients seen in the PED each year, approximately 85% of patients are discharged with a prescription for medication. This makes the PED an ideal setting to implement a health literacy intervention to reduce medication administration errors at home. The investigators are proposing to conduct a randomized controlled trial of an educational module focused on how to administer antibiotics at home and test whether there is an improvement in care practices.

ELIGIBILITY:
Inclusion Criteria:

Caregivers of:

* Patients aged 2 months to 8 years
* Patients triaged to Emergency Severity Index (ESI) level 4 or 5 in the pediatric emergency department.
* Patients with at least one prescription for a liquid, tablet or ointment antibiotic.

Exclusion Criteria:

Caregivers of:

* Patients in need of immediate care.
* Patients hospitalized.

Ages: 2 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Score on the telephone interview post-test | 48-72 hours post Emergency Department visit
  Subject scores will be dichotomized in the follow way: anything less than 100% will be considered incorrect, a score of 100% will be considered correct.

SECONDARY OUTCOMES:
Prevalence of perfect performance on each element of the questionnaire | 48-72 hours post Emergency Department visit
  Each answer on the telephone interview post-test will be dichotomized into a correct/incorrect answer.

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Subramony, MD, MBA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States